CLINICAL TRIAL: NCT05660811
Title: Optimal Antiplatelet Treatment to Achieve Stroke Avoidance and Fall in Bleeding Events Following Left Atrial Appendage Closure - Chronic Kidney Disease (SAFE LAAC CKD). Comparative Health Effectiveness Ancillary Study - PILOT
Brief Title: Optimal Antiplatelet Therapy Following Left Atrial Appendage Closure in Dialyzed Patients
Acronym: SAFE LAAC CKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKD/1458/21
Record Dates: First submitted 2022-07-15; First posted 2022-12-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; stroke; bleeding; left atrial appendage; dialysis
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Long-Term Care; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30 days DAPT and long-term treatment with a single antiplatelet agent (Other): short postimplantation dual antiplatelet therapy and long-term treatment with a single antiplatelet agent
  Interventions: Drug: short postimplantation dual antiplatelet therapy; Drug: long-term treatment with a single antiplatelet agent
- 6 months DAPT and long-term treatment with a single antiplatelet agent (Other): extended postimplantation dual antiplatelet therapy and long-term treatment with a single antiplatelet agent
  Interventions: Drug: extended postimplantation dual antiplatelet therapy; Drug: long-term treatment with a single antiplatelet agent
- 30 days DAPT and 6 months treatment with a single antiplatelet agent (Other): short postimplantation dual antiplatelet therapy and 6 months treatment with a single antiplatelet agent
  Interventions: Drug: short postimplantation dual antiplatelet therapy; Drug: 6 months treatment with a single antiplatelet agent
- 6 months DAPT and 6 months treatment with a single antiplatelet agent (Other): extended postimplantation dual antiplatelet therapy and 6 months treatment with a single antiplatelet agent
  Interventions: Drug: extended postimplantation dual antiplatelet therapy; Drug: 6 months treatment with a single antiplatelet agent

INTERVENTIONS:
Drug: short postimplantation dual antiplatelet therapy — continuing dual antiplatelet therapy up until 6 months after left atrial appendage occlusion with Amplatzer Amulet
  Arms: 30 days DAPT and 6 months treatment with a single antiplatelet agent; 30 days DAPT and long-term treatment with a single antiplatelet agent
Drug: extended postimplantation dual antiplatelet therapy — stopping dual antiplatelet therapy after 30 days after left atrial appendage occlusion with Amplatzer Amulet and continuing single antiplatelet agent up until 6 months
  Arms: 6 months DAPT and 6 months treatment with a single antiplatelet agent; 6 months DAPT and long-term treatment with a single antiplatelet agent
Drug: long-term treatment with a single antiplatelet agent — continuing long-term treatment with single antiplatelet agent
  Arms: 30 days DAPT and long-term treatment with a single antiplatelet agent; 6 months DAPT and long-term treatment with a single antiplatelet agent
Drug: 6 months treatment with a single antiplatelet agent — continuing single antiplatelet agent up until 6 months
  Arms: 30 days DAPT and 6 months treatment with a single antiplatelet agent; 6 months DAPT and 6 months treatment with a single antiplatelet agent

SUMMARY:
SAFE-LAAC CKD Trial has been designed to gather data on the most optimal strategy of antiplatelet therapy after transcatheter left atrial appendage occlusion with Amplatzer or WATCHMAN device in patients with the end-stage renal disease treated with chronic haemodialysis or peritoneal dialysis

DETAILED DESCRIPTION:
Background:

Transcatheter left atrial appendage closure (LAAC) has been shown to be non-inferior to oral anticoagulation in preventing cardioembolic strokes associated with atrial fibrillation. However, an optimal antithrombotic treatment regimen following successful LAAC remains an unresolved issue and may significantly contribute to long-term safety and efficacy. Nowadays LAAC is mainly performed in patients with contraindications for oral anticoagulation due to high bleeding risk. Dialyzed patients with end-stage renal disease and atrial fibrillation have simultaneously high thromboembolic and bleeding risk. Such patients were excluded from randomized trials and data on the LAAC efficacy in this population is limited thus prospective studies are warranted.

Objective:

SAFE-LAAC CKD Trial has been designed as a comparative health effectiveness study with the following aims:

1. compare the safety and efficacy of 30 days vs. 6 months of dual antiplatelet therapy following LAAC with Amplatzer or WATCHMAN device (randomized comparison)
2. compare the safety and efficacy of stopping all antithrombotic and antiplatelet agents 6 months after LAAC vs. long-term treatment with a single antiplatelet agent (nonrandomized comparison)

Patient population:

Patients (n=80) with the end-stage renal disease treated with chronic haemodialysis or peritoneal dialysis, after successful LAAC with Amplatzer or WATCHMAN device

Perspective:

Results of this pilot trial will provide: 1. data to aid practitioners and guideline writers recommend the most optimal antithrombotic treatment after LAAC, 2. data on the safety and efficacy of LAAC in dialyzed patients, and 3. data to support power calculations for designing future randomized trials.

Methodology:

SAFE LAAC CKD has been designed as a multicenter (planned contribution of 7 centers in Poland), open-label, comparative health effectiveness trial with central, independent adjudication of events comprising the primary end-point. The first part of the trial is randomized and after 6 months of follow-up continues for another 12 months as a non-randomized study.

Timeline:

The duration of the trial has been planned for 5 years. The enrollment phase has been planned for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Successful left atrial appendage occlusion with Amplatzer or WATCHMAN device within 37 days prior to randomization
* End-stage renal disease treated with chronic haemodialysis or peritoneal dialysis
* Participant's age 18 years or older at the time of signing the informed consent form
* Participant is willing to follow all study procedures; especially the randomized antiplatelet treatment regimen
* Participant is willing to sign the study informed consent form

Exclusion Criteria:

* Indications to dual antiplatelet therapy other than left atrial appendage occlusion at the time of enrollment and/or predicted appearance of such indications within the duration of the trial (e.g. planned coronary revascularization)
* Indications to anticoagulation at the time of enrollment and/or predicted appearance of such indications within the duration of the trial (e.g. pulmonary embolism). Does not apply to anticoagulation used during dialysis
* Known allergy to clopidogrel and/or acetylsalicylic acid precluding its administration as specified by the protocol
* Peridevice leak >5mm on imaging study preceding enrollment
* Left atrial thrombus on an imaging study performed after successful left atrial appendage closure but before enrollment
* Life expectancy of fewer than 18 months
* Participation in other clinical studies with experimental therapies at the time of enrollment and/or preceding 3 months
* Women who are pregnant or breastfeeding; women of childbearing potential who do not consent to apply at least two methods of contraception. This criterion does not apply to women 2 years post menopause (with a negative pregnancy test 24 hours before randomization if <55 years old) or after surgical sterilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy (a composite of ischemic stroke, transient ischaemic attack, peripheral embolism, nonfatal myocardial infarction, cardiovascular mortality, all-cause mortality, left atrial appendage thrombus) | 17 months
  Event rates reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Safety (moderate and/or severe bleeding (BARC type 2, 3, and 5) | 17 months
  Event rates reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);

SECONDARY OUTCOMES:
Ischemic stroke | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Transient ischaemic attack | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Peripheral embolism | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Nonfatal myocardial infarction | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Cardiovascular mortality | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
All-cause mortality | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Moderate and/or severe bleeding (BARC type 2,3, and 5) | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Left atrial appendage thrombus | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Any bleeding | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
New moderate or major (≥4 mm) ischemic brain lesions on magnetic resonance imaging | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Change in cognition score as detected by the Addenbrooke's cognitive examination (ACE-III) | 17 months
  ACE-III is a screening test that is composed of tests of attention, orientation, memory, language, visual perceptual, and visuospatial skills. The total range of raw score is 0-100. A higher score indicates more intact cognitive functioning.
Dialysis access thrombosis | 17 months
  Event rate reported per 100 patient-years (calculated as 100*Number of Participants with events/Total patient-years);
Safety and efficacy of the procedure in the periprocedural period and 1-month follow-up based on registry data | 1-month
  1-month event rate of: cardiac arrest, device embolism, tamponade, pericardial effusion, stroke/TIA/myocardial infarction/peripheral embolus, access site bleeding/vascular complications, bleeding complications unrelated to access site (Number of Participants with event/Total patient number)

OTHER OUTCOMES:
Number of new ischemic brain lesions on magnetic resonance imaging | 17 months
Volume of new ischemic brain lesions on magnetic resonance imaging | 17 months
The change from baseline in the cumulative dose of heparin anticoagulation used during haemodialysis | 17 months
The change from baseline in the dose of erythropoietin used | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Pracon, MD PhD, Principal Investigator — Coronary and Structural Heart Diseases Department, National Institute of Cardiology, Warsaw, Poland
Locations (1):
- National Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided